CLINICAL TRIAL: NCT06508879
Title: Randomized Controlled Trial: Does the Use of Occlusive Hydrocolloid Silver-containing Wound Dressing After Sternotomy Reduce Surgical Side Infection After Cardiac Surgery?
Brief Title: Does Occlusive Hydrocolloid Silver-containing Wound Dressing After Sternotomy Reduce Surgical Side Infection After Cardiac Surgery?
Acronym: OHSCWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Mainz (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Dr. med. Kathrin Dohle, Cardiac surgery specialist, University Medical Center Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OHSCWD for sternotomy
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Surgical Site Infection; Cardiac Surgery; Advanced Dressing; Postoperative Care
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study was designed as a single-center randomized controlled trial. Primary endpoint was overall rate of incidence of any kind of SSI. Secondary endpoints were number of dressing changes, severity of SSI and need for treatment. Wounds were monitored daily until the 7th and on the 30th postoperative day.
Masking Description: The patients were blinded until the time of the intervention (application of the bandage after surgery). Due to the nature of this study, it was not possible to conceal the treatment after the procedure, as patients could see their bandages and find out their allocation. Using methods to conceal the dressings (covering with neutral dressing) would have changed the nature of the dressings and affected the treatment. The study team could also see the bandages and was therefore not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): a standard wound dressing composed of sterile gauze and adhesive tape was applied under sterile conditions. In the absence of bleeding, excessive wound secretion, or detachment, the dressing was left on the wound until the second postoperative day (POD 2), otherwise, it was changed immediately. Starting at POD 2, the dressing was changed daily under aseptic conditions until the wound remained dry (between POD 3-5). In the absence of bleeding, excessive wound secretion, or detachment, the wound was then left uncovered. This practice corresponded to the standard treatment of cardiothoracic patients in our department at the time of initiating this study.
  Interventions: Other: Standard Care (sterile gauze and adhesive tape)
- Test Group (Experimental): directly after closing the wound, an occlusive hydrocolloid silver-containing wound dressing (Aquacel Ag Surgical®, ConvaTec, Oklahoma City, OK, USA) was applied under sterile conditions and, in the absence of bleeding; excessive wound secretion, or detachment, was maintained on the wound until POD 5, at which time the dressing was removed. In case of bleeding, excessive wound secretion, or detachment, the dressing was removed, the wound was cleaned, and a new sterile hydrocolloid wound dressing applied under aseptic conditions.
  Interventions: Combination Product: Aquacel Ag Surgical®

INTERVENTIONS:
Combination Product: Aquacel Ag Surgical® — Presurgical preparation was identical in both groups and no further intervention in patient treatment was made. See descpription of arms.
  Arms: Test Group
Other: Standard Care (sterile gauze and adhesive tape) — Presurgical preparation was identical in both groups and no further intervention in patient treatment was made. See descpription of arms.
  Arms: Control Group

SUMMARY:
Wound healing disorders are a major problem in cardiac surgery. They prolong the inpatient stay and are associated with a high health and, above all, psychological burden for patients. They also represent a major organizational, medical and financial challenge for the treatment team. There is therefore still a great need for effective prevention of wound healing disorders. It goes without saying that wound management plays a major role in the development of wound healing disorders. Nowadays, there are a large number of products from various manufacturers and studies for efficient wound healing disorder prophylaxis. One point of criticism is that most of the existing studies are financed by the manufacturer. Due to the otherwise broad range of applications for all wounds in various specialist areas, it remains to be clarified whether such products can achieve a reduction in the rate of wound healing disorders, especially in cardiac surgery. After extensive literature research, we are of the opinion that the Aquacel Surgical Ag dressing, a new silver-coated hydrocolloid dressing, can be offered to cardiac surgery patients at our clinic as an effective prophylaxis against wound healing disorders.The study is a randomized prospective clinical trial. It is being conducted at the Clinic for Cardiothoracic and Vascular Surgery and has already been approved by the Rhineland-Palatinate Ethics Committee. The study should include 440 heart patients and last for 12 months. It will compare the Aquacel Surgical Ag bandage against our conventional methods. This study is being conducted independently of the industry. We want to prove that an intelligent investment in the prophylaxis of wound healing disorders is worthwhile for both patients and the clinic. If the outcome of the study is positive, this dressing will be be used regularly in our cardiac surgery clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary artery bypass surgery
2. Elective and primary surgery (no reoperations)
3. Complete median sternotomy
4. Age under 90 years
5. Weight in the range of 50-140kg
6. No known allergy to silver or other wound dressings
7. No immunosuppressive therapy or hormonal substitution therapy, except for thyroid hormone
8. Capacity to consent

Exclusion Criteria:

1. Failure of medical personnel to adhere to study protocol, e.g., not applying the right wound dressing according to study protocol
2. Patients own decision
3. Lack of harvesting of at least one internal thoracic artery
4. Peri- and post-operative ventilation for >48h
5. Re-thoracotomy for reasons other than SSI, e.g., bleeding
6. Mortality within the first 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
SSI rate | 30 days
  overall rate of incidence of any kind of SSI

SECONDARY OUTCOMES:
dressing changes | 7 days
severity of SSI | 30 days
need for treatment | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Surgery, University Hospital of Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No